CLINICAL TRIAL: NCT02430974
Title: Icotinib as Maintenance Treatment After Chemotherapy for Patients Undergoing Resection of EGRF Mutation-positive Non-small Cell Lung Cancer
Brief Title: Chemotherapy of NSCLC With or Without Icotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFYYXWK-CKC1102
Record Dates: First submitted 2015-04-26; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

ARMS (2):
- Chemotherapy (No Intervention): patients received four cycles of platinum-based doublet chemotherapy (150 mg/m2 paclitaxel plus 80 mg/m2 nedaplatin or 30mg/m2 lobaplatin on day one of a three-week cycle).
- Chemotherapy & Icotinib (Experimental): patients received four cycles of platinum-based doublet chemotherapy (150 mg/m2 paclitaxel plus 80 mg/m2 nedaplatin or 30mg/m2 lobaplatin on day one of a three-week cycle).Two weeks after chemotherapy completed, patients assigned to the consolidation therapy group began oral icotinib treatment (125 mg, thrice daily). Icotinib treatment continued for four to eight months, or until the occurrence of disease relapse, metastasis or unacceptable icotinib or chemotherapy toxicity.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Patients in experimental group will receive oral Icotinib for 4-8months.
  Arms: Chemotherapy & Icotinib

SUMMARY:
Epidermal growth factor receptor (EGFR) mutations occur in up to 50% of Asian patients with non-small cell lung cancer (NSCLC). Treatment of advanced NSCLC patients with EGFR-tyrosine kinase inhibitors (EGFR-TKI) confers a significant survival benefit. This study assessed the efficacy and safety of chemotherapy with or without icotinib in patients undergoing resection of stage IB to IIIA EGFR-mutated NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing completely resection of EGRF mutation-positive NSCLC
* Staging ⅠB (with high risk factor) to ⅢA
* PS = 0 or 1
* Adequate hematological, biochemical and organ functions

Exclusion Criteria:

* Systemic anticancer therapy prior to surgery, other malignancies before or during the study, any unstable illness, women who were pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | from the date of surgery until the date of first confirmed disease relapse or metastasis, assessed up to 5 years

SECONDARY OUTCOMES:
Number of Participants with Adverse Effects | duration of receiving chemotherapy and oral icotinib, expected to be 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kaican Cai, MD, Principal Investigator — Nanfang Hospital, Southern Medical University

REFERENCES:
- [Derived] Feng S, Wang Y, Cai K, Wu H, Xiong G, Wang H, Zhang Z. Randomized Adjuvant Chemotherapy of EGFR-Mutated Non-Small Cell Lung Cancer Patients with or without Icotinib Consolidation Therapy. PLoS One. 2015 Oct 16;10(10):e0140794. doi: 10.1371/journal.pone.0140794. eCollection 2015. PMID 26474174